CLINICAL TRIAL: NCT04045756
Title: Short-term Efficacy of Transperineal Laser Ablation (TPLA) With Image Fusion and Multi-parametric (mpMRI) Follow-up in Focal Low-intermediate Risk Prostate Cancer: Interventional Pilot Study
Brief Title: Focal Laser Ablation for the Treatment of Focal Low-Intermediate Risk Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Guglielmo Manenti, Principal Investigator, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.S. 68.19
Record Dates: First submitted 2019-07-11; First posted 2019-08-06 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; laser ablation; mpMRI; interventional radiology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ECHOLASER X4 Socratelite (Experimental): Optic fiber of 300um will be inserted at a distance of 8-10mm from the urethra. Each ablation lasts 6 minutes. Each fiber ablates at an energy of 1800J with a power of 2-3W. Treatment lasts for about 30 minutes.
  Interventions: Device: Procedure/Surgery: Transperineal Focal Laser Ablation (TPLA)

INTERVENTIONS:
Device: Procedure/Surgery: Transperineal Focal Laser Ablation (TPLA) — The intervention will take place in an ambulatory setting of the interventional radiology department using the combined Echolaser XVG system. The treatment consists of a local anesthesia to the perineal region. Within each needle, an optic fiber of 300um will be inserted. Each ablation lasts 6 minutes and each fiber ablates 1800J at a power of 2-3W. At the end of the ablation there is a pull-back of about 1cm from the original ablation location. According to the dimension of the middle lobe of the prostate, multiple pullbacks can be used. The total ablation is 3600J for 2 fibers (1800J/ fiber) at the power of 2-3W for a total duration of about 30minutes. At the end of the treatment, a 20mg bollous of i.v. corticosteriods () is given for anti-edema and anti-inflammatory effects. Antibiotic therapy (Cirpofloxacin 500mg and gastroprotective therapy is given for 5 days. After an adequate amount of time for observation, the patient is dismissed.

SUMMARY:
Short-term Efficacy of Transperineal Laser Ablation (TPLA) with Image Fusion and Multi-parametric (mpMRI) Follow-up in Focal Low-intermediate Risk Prostate Cancer. It is an interventional pilot study. The clinical evaluation will be carried out at different times as follows:

Time 0: recruitment and eligibility assessment (patient selection) Time 1: interview, signing of informed consent and enrollment Time 2: FLA treatment and control with multiparametric MRI of the post-procedural prostate.

Time 3-4-5-6: follow up to 1 (T3), 6 (T4), 12 (T5) and 24 (T6) months from the procedure.

The primary objective of the study is to evaluate the short-term (2 years) efficacy of FLA treatment of low-intermediate risk prostate cancer Secondary objective is to investigate multiparametric prostate MRI as a follow-up diagnostic investigation, evaluating possible glandular morphostructural changes and their correlation with clinical data.

DETAILED DESCRIPTION:
Short-term Efficacy of Transperineal Laser Ablation (TPLA) With Image Fusion and Multi-parametric (mpMRI) Follow-up in Focal Low-intermediate Risk Prostate Cancer. It is an interventional pilot study.

The recruitment and evaluation of eligibility will be done by the Multidisciplinary Neoplasms Group of the Uro-Genital System, already operating within the Tor Vergata Polyclinic Foundation and formed by the following Operating Units:

UOSD Urology, UOC Diagnostic Imaging, UOC Medical Oncology, UOC Radiotherapy, UOSD Pathological Anatomy, UOC Nuclear Medicine. The Multidisciplinary Group will propose and evaluate patients that can be recruited based on inclusion and exclusion criteria. The patient considered eligible for the study will be adequately informed by the UOSD Urology / UOC Diagnostic Imaging regarding the therapeutic possibilities for the specific disease stage.

If the patient expresses an interest in participating in the study, he will be given informed consent.

Once the informed consent has been signed, the patient will be considered enrolled in the study.

Pre-procedural evaluation

Pre-treatment clinical-instrumental-blood chemistry tests include:

* Electrocardiogram
* Complete blood count, blood ureanitrogen (BUN), creatinine, sodium, potassium, coagulation tests
* Urine examination and urine culture
* Evaluation of the post-voiding residue
* Uroflowmetry (if IPSS> 7)

Questionnaires:

* IPSS-QoL
* IIEF

Focal laser ablation treatment (FLA):

The treatments will be performed by the Diagnostic Imaging team, on a Day Hospital basis, using the combined Echolaser XVG system (Elesta s.r.l - Calenzano (FI)).

The EchoLaser Therapy is a micro-invasive percutaneous procedure that uses the laser light transmitted through applicators (optical fibers) for a few minutes, causing the affected tissue to warm up until it is irreversibly damaged in "situ", without the need to remove it.

All this thanks to the combined action of an increase in the local temperature and the exposure time. The interaction of laser radiation with a wavelength of 1064nm (in the range of the therapeutic window) is excellent, with low radiation absorption and excellent light penetration. The laser light is conveyed from the source to the fabric through extremely flexible, small-caliber (300 micron diameter) flat-tip quartz optical fibers, introduced percutaneously by thin needles (21 Gauge).

The EchoLaser Therapy, through flat-tipped fibers, produces an ellipsoidal coagulation area (an area where the tissue has irreversible damage). A possible multi-fiber approach can extend the coagulation area.

The EchoLaser Therapy can be performed under ultrasound guidance for real-time monitoring of the correct positioning of the laser light applicators and the effective extension of the damage to the tumor lesion.

The procedure will be performed with a patient in a lithotomy position and in safe conditions according to the current legislation for treatments with laser systems (such as protective glasses).

Treatment includes local anesthesia of the perineal region, under ultrasound guidance. At the discretion of the medical team, intravenous sedation can be performed.

1-2 spinal needles 21G will be inserted into the intralesional site by ultrasound-guided transperineal route after MRI / TRUS image fusion. In each needle a 300 micron optical fiber will be inserted (Elesta s.r.l., Calenzano (FI)). For each lighting, for about 6 minutes, a maximum energy of 1800 J per fiber will be delivered, with a power of 2-5 Watts. If necessary, the needle and fiber will be retracted for about 1 cm ("pull-back"). Further lighting will follow, with delivery and duration and power equal to the previous one.

Immediately after the procedure, the patient will be asked to complete the VAS score for the assessment of pain felt during the procedure.

Complications: The potential complications of the FLA technique are:

* Peri-operative: perineal and hypogastric pain, perineal hematoma, hematuria, acute urinary retention, fever, dysuria
* Postoperative: perineal pain, LUTS, persistent hematuria, hematospermia, erectile dysfunction, urinary incontinence Complications will be investigated prospectively using the Clavien-Dindo classification

Follow-up: The clinical evaluation will be carried out at different times:

Post procedural follow up A multi-parametric prostate MRI will be performed immediately after the treatment. At the end of the treatment the resumption of spontaneous diuresis will be checked and in the case of acute urinary retention / clinically significant hematuria a bladder catheter will be inserted.

An oral cortisone drug (Deflazacort 30 mg) or other anti-edema therapy will be prescribed if specifically contraindicated by the patient.

Any complications will be recorded according to the Clavien-Dindo classification The patient will be discharged with antibiotic therapy, pain relief when needed and gastroprotective for 5-7 days.

Patients will receive a telephone contact to use to communicate any post-operative emergencies.

Post-discharge follow-up The specialist follow-up visit to 1 (T3), 6 (T4), 12 (T5) and 24 (T6) months from the procedure will be conducted by the UOSD Urology.

Any reported complications will be recorded according to the Clavien-Dindo classification.

The patient will be asked to complete the IPSS-QoL and IIEF questionnaires and will view the total serum PSA (T4-T5-T6).

Multi-parametric prostate MRI will be performed at T4-T6. Transperineal prostatic control biopsy will be performed with fusion target (ablated zone) and systematic technique (T4-T6).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Over 45 years old
* Prostate cancer identified after prostatic biopsy with fusion of images with target and systematic samples (> 12)
* Intermediate progression risk (Gleason Score 3 + 4 or 4 + 3; PSA <15 ng / ml; clinical stage T1-T2a)
* Low risk of progression (Gleason score 3 + 3) only in patients who wish to leave or who refuse the active surveillance protocol and who refuse validated treatments for the treatment of organo-confined prostate cancer: radical surgery and / or radiotherapy

Exclusion Criteria:

* Prostate cancer Gleason Score> = 4 + 4.
* Clinical stage> T2a
* PSA> 15 ng / ml
* Presence of metastases from prostate lymph node, bone or visceral carcinoma detected by bone scintigraphy, total body CT or PET-CT
* Serious coagulation disorders not correctable
* Unavailable or replaceable anticoagulant and / or antiplatelet therapy
* Inadequate compliance
* Presence of pacemakers
* Contraindications to MRI (claustrophobia, ear implants, metal prostheses)
* Paramagnetic contrast agent allergy
* Acute and / or chronic renal failure (GFR <50 mL / min and serum creatinine> 1.5 mg / dl)
* Tumor volume <15 ml measured on MRI

Ages: 46 Years to 86 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-08-02 (Estimated); Study Completion 2024-08-02 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  Cancer control defined as the percentage of patients with disease free survival according to the pathological MR-guided biopsy results in a 5 year period.
Evaluation of Complications of prostate Laser Ablation on the Treatment of Focal Low-Intermediate Risk Prostate Cancer by use of mp-MRI. | 5 years
  Evaluation of the post-procedural complications by mpMRI. In particular damage to neuro-vascular bundles, seminal vescicles and peri-prostatic fat will be checked.

SECONDARY OUTCOMES:
Reproducibility of mpMRI in correlation with biopsy in order to establish positive/negative predictive diagnostic values of MRI in residual/relapsing tumors | 5 years
  Evaluation of multi-parametric MRI of the prostate and evaluate the response to focal laser ablation treatment for focal low-intermediate prostate cancer by biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Manenti, MD PhD, Principal Investigator — Fondazione Policlinico Tor Vergata
Locations (1):
- Policlinico Tor Vergata (PTV) Foundation: Department di Biomedicine and Prevention, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
Create an international registry to assess long-term effectiveness of transperineal laser ablation for focal prostate cancer, to assess functional outcomes, to assess safety, to determine baseline patient characteristics, to collect information on possible differences between centres applying treatment of transperineal laser ablation and to explore the optimal treatment indications and possible limitations. It an international prospective observational registry in which data is recorded of patients who are treated with transperineal laser ablation for low-intermediate risk focal prostate cancer.
Supporting Information: Study Protocol, ICF
Time Frame: This registry will be open for inclusion for five years. Since individual patients will have a follow-up of five years, the total study duration will be 10 years.
Access Criteria: Every accredited centre that performs TPLA procedures, wants to participate and signs the regulatory document and obtains ethical committee approval can participate
URL: https://www.flaprostate.com/

REFERENCES:
- [Background] Patelli G, Ranieri A, Paganelli A, Mauri G, Pacella CM. Transperineal Laser Ablation for Percutaneous Treatment of Benign Prostatic Hyperplasia: A Feasibility Study. Cardiovasc Intervent Radiol. 2017 Sep;40(9):1440-1446. doi: 10.1007/s00270-017-1662-9. Epub 2017 May 4. PMID 28474112
- [Background] Lindner U, Lawrentschuk N, Trachtenberg J. Image guidance for focal therapy of prostate cancer. World J Urol. 2010 Dec;28(6):727-34. doi: 10.1007/s00345-010-0604-9. Epub 2010 Oct 21. PMID 20963422
- [Background] Lindner U, Weersink RA, Haider MA, Gertner MR, Davidson SR, Atri M, Wilson BC, Fenster A, Trachtenberg J. Image guided photothermal focal therapy for localized prostate cancer: phase I trial. J Urol. 2009 Oct;182(4):1371-7. doi: 10.1016/j.juro.2009.06.035. Epub 2009 Aug 14. PMID 19683262
- [Background] Goldberg SN, Grassi CJ, Cardella JF, Charboneau JW, Dodd GD 3rd, Dupuy DE, Gervais D, Gillams AR, Kane RA, Lee FT Jr, Livraghi T, McGahan J, Phillips DA, Rhim H, Silverman SG; Society of Interventional Radiology Technology Assessment Committee. Image-guided tumor ablation: standardization of terminology and reporting criteria. J Vasc Interv Radiol. 2005 Jun;16(6):765-78. doi: 10.1097/01.RVI.0000170858.46668.65. PMID 15947040
- [Background] Bremer C, Kreft G, Roggan A, Filler T, Reimer P. Ex vivo evaluation of novel miniaturized laser-induced interstitial thermotherapy applicators for effective small-volume tissue ablation. Invest Radiol. 2001 Jun;36(6):327-34. doi: 10.1097/00004424-200106000-00005. PMID 11410753
- [Background] Costello AJ, Johnson DE, Bolton DM. Nd:YAG laser ablation of the prostate as a treatment for benign prostatic hypertrophy. Lasers Surg Med. 1992;12(2):121-4. doi: 10.1002/lsm.1900120202. PMID 1374142
- [Background] Oto A, Sethi I, Karczmar G, McNichols R, Ivancevic MK, Stadler WM, Watson S, Eggener S. MR imaging-guided focal laser ablation for prostate cancer: phase I trial. Radiology. 2013 Jun;267(3):932-40. doi: 10.1148/radiol.13121652. Epub 2013 Feb 25. PMID 23440319
- [Background] van Luijtelaar A, Greenwood BM, Ahmed HU, Barqawi AB, Barret E, Bomers JGR, Brausi MA, Choyke PL, Cooperberg MR, Eggener S, Feller JF, Frauscher F, George AK, Hindley RG, Jenniskens SFM, Klotz L, Kovacs G, Lindner U, Loeb S, Margolis DJ, Marks LS, May S, Mcclure TD, Montironi R, Nour SG, Oto A, Polascik TJ, Rastinehad AR, De Reyke TM, Reijnen JS, de la Rosette JJMCH, Sedelaar JPM, Sperling DS, Walser EM, Ward JF, Villers A, Ghai S, Futterer JJ. Focal laser ablation as clinical treatment of prostate cancer: report from a Delphi consensus project. World J Urol. 2019 Oct;37(10):2147-2153. doi: 10.1007/s00345-019-02636-7. Epub 2019 Jan 22. PMID 30671638
- [Background] Walser E, Nance A, Ynalvez L, Yong S, Aoughsten JS, Eyzaguirre EJ, Williams SB. Focal Laser Ablation of Prostate Cancer: Results in 120 Patients with Low- to Intermediate-Risk Disease. J Vasc Interv Radiol. 2019 Mar;30(3):401-409.e2. doi: 10.1016/j.jvir.2018.09.016. PMID 30819483
- [Background] Lepor H. Vascular targeted photodynamic therapy for localized prostate cancer. Rev Urol. 2008 Fall;10(4):254-61. PMID 19145269
- [Derived] Manenti G, Perretta T, Nezzo M, Fraioli FR, Carreri B, Gigliotti PE, Micillo A, Malizia A, Di Giovanni D, Ryan CP, Garaci FG. Transperineal Laser Ablation (TPLA) Treatment of Focal Low-Intermediate Risk Prostate Cancer. Cancers (Basel). 2024 Apr 3;16(7):1404. doi: 10.3390/cancers16071404. PMID 38611082

DOCUMENTS (2):
  • Informed Consent Form (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT04045756/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04045756/Prot_SAP_001.pdf